CLINICAL TRIAL: NCT04576481
Title: Literary Promotion Using Automated Hovering to Improve Development in Young Low-Income Children
Brief Title: Literacy Promotion Using Automated Hovering
Acronym: LP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 19-017199
Record Dates: First submitted 2020-09-25; First posted 2020-10-06 (Actual); Results first posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-09

CONDITIONS: Parent-Child Relations; Parenting; Literacy
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Intervention Model Description: The intervention consists of 3 intervention groups. Participants will be stratified by site and randomized 1:1:1 to receive one of the 3 AH interventions for an 8-week duration.
Who Masked: Outcomes Assessor
Masking Description: Participants will not be blinded to their treatment assignment. However, research staff will be blinded to treatment assignment when collecting study data.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Texting (Active Comparator): Consist of daily text messages on shared reading
  Interventions: Behavioral: Texting
- Group 2: Regret (Experimental): Will consist of Group 1 plus social comparisons.
  Interventions: Behavioral: Texting; Behavioral: Regret
- Group 3: Lottery (Experimental): Will consist of Group 2 plus availability of a weekly lottery.
  Interventions: Behavioral: Texting; Behavioral: Regret; Behavioral: Lottery

INTERVENTIONS:
Behavioral: Texting — Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
Behavioral: Regret — Personalized coaching content will be made available to participants through links in the text messages and will provide comparisons of their reading frequency with that of other participants.
  Arms: Group 2: Regret; Group 3: Lottery
Behavioral: Lottery — Participants who reply to a text message that they read on a particular day will be entered into daily and weekly drawings to receive cash payments.
  Arms: Group 3: Lottery

SUMMARY:
The purpose of this study is to incorporate behavioral economics (BE) approaches to determine whether 3 novel interventions of varying intensity improve the frequency of parent-child reading behaviors among low-income families. In the first phase, 10 parents will be recruited to participate in rapid cycle interviews to determine the appropriateness of text messages. In the second phase, 45 participants will be randomized to comparative groups to test the effects of automated hovering and other BE approaches on frequency of parent-child shared reading. Investigators long-term goal is to test the effects of these approaches to promote child language and socio-emotional development.

DETAILED DESCRIPTION:
Early childhood is a sensitive period in which young children develop language and socio-emotional skills foundational for school readiness. Unfortunately, poor vulnerable children experience disparities in these critical areas of development. Parent-child shared reading can help ameliorate these disparities, yet low-income parents do not consistently engage in this activity. Behavioral economics approaches utilizing automated hovering (AH) have the potential to increase parent-child shared reading through text messages and financial inducements.

The study design is a two-phase study consisting of a qualitative component followed by a prospective, randomized comparative group trial to test the effects of AH approaches to increase parent-child shared reading. A total of 55 eligible children and their parents will be recruited from participating practices to achieve a diverse sample of children.

In the first phase, 10 parents will be recruited to participate in brief rapid cycle interviews to assess the appropriateness of text message reminders. In the second phase, forty-five participants will be randomized 1:1:1 to receive one of the 3 AH interventions: 1) daily text message reminders (texting), 2) daily text message reminders with social comparisons (regret) or 3) daily text message reminders with social comparisons and weekly lottery entries (lottery). All interventions are related to principles of behavioral economics in order to provide external motivation. There will be 15 participants per group to adequately assess feasibility and acceptability, the primary outcome.

Descriptive statistics for demographic, home reading environment, and parenting stress measured at baseline will be examined across the three groups to assess the success of the randomization. To assess feasibility and acceptability, Investigators will assess the proportion of participants who receive and report a daily reading behavior each week across all groups, the proportion of participants who access coaching content in group 2 & 3, and the proportion of participants who participate in the weekly lottery in group 3, and satisfaction scores in all groups. Secondary outcomes including differences between groups in weekly reading frequency, home reading environment, and child socio-emotional scores between groups will be assessed using standard inferential statistics and intention-to-treat analysis.

The results of this study may assist health care providers and researchers in testing the feasibility of AH approaches to improve parent-child shared reading and prepare for a larger efficacy trial.

ELIGIBILITY:
Inclusion Criteria:

* Parents who:

  * Have an infant aged 6-24 months
  * Have access to a smart phone with text messaging capabilities
  * Have completed an informed consent
* Children who:

  * Are aged 6-24 months old

Exclusion Criteria:

* Parents who:

  - Non-English speaking
* Children who:

  * Were born premature (estimated gestational age < 35 weeks)
  * Have been diagnosed with congenital malformations or genetic syndromes which place them at risk for developmental delays

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 55 (Actual)
Dates: Start 2020-11-17 (Actual); Primary Completion 2022-02-04 (Actual); Study Completion 2022-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Guevara, MD, MPH, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
A complete, cleaned, and de-identified dataset will be made available to other investigators after all analyses have been conducted and within twelve months of the end of the final year of funding to allow for publication of all study aims. To obtain this data set, other investigators will need to contact the study Principal Investigator (PI) who will provide a data sharing agreement. The data sharing agreement will permit a deidentified data set to be shared once an Institutional Review Board (IRB) protocol has been approved at the investigators' home institution and the investigators have signed a pledge to not attempt to identify individual study subjects. The data set will be made available on a Compact Disc Read-Only Memory (CD-ROM) or through a secure File Transfer Protocol (FTP) site.
Supporting Information: Study Protocol, SAP
Time Frame: 12 months after the end of the final year of funding.
Access Criteria: REDCap access

REFERENCES:
- [Background] National Research Council (US) and Institute of Medicine (US) Committee on Integrating the Science of Early Childhood Development; Shonkoff JP, Phillips DA, editors. From Neurons to Neighborhoods: The Science of Early Childhood Development. Washington (DC): National Academies Press (US); 2000. Available from http://www.ncbi.nlm.nih.gov/books/NBK225557/ PMID 25077268
- [Background] Rosenberg SA, Zhang D, Robinson CC. Prevalence of developmental delays and participation in early intervention services for young children. Pediatrics. 2008 Jun;121(6):e1503-9. doi: 10.1542/peds.2007-1680. Epub 2008 May 26. PMID 18504295
- [Background] Blair C, Raver CC. Poverty, Stress, and Brain Development: New Directions for Prevention and Intervention. Acad Pediatr. 2016 Apr;16(3 Suppl):S30-6. doi: 10.1016/j.acap.2016.01.010. PMID 27044699
- [Background] The pediatrician's role in development and implementation of an Individual Education Plan (IEP) and/or an Individual Family Service Plan (IFSP). American Academy of Pediatrics. Committee on Children with Disabilities. Pediatrics. 1999 Jul;104(1 Pt 1):124-7. doi: 10.1542/peds.104.1.124. PMID 10390275
- [Background] Centers for Disease Control and Prevention (CDC). Economic costs associated with mental retardation, cerebral palsy, hearing loss, and vision impairment--United States, 2003. MMWR Morb Mortal Wkly Rep. 2004 Jan 30;53(3):57-9. PMID 14749614
- [Background] Cates CB, Dreyer BP, Berkule SB, White LJ, Arevalo JA, Mendelsohn AL. Infant communication and subsequent language development in children from low-income families: the role of early cognitive stimulation. J Dev Behav Pediatr. 2012 Sep;33(7):577-85. doi: 10.1097/DBP.0b013e318264c10f. PMID 22947884
- [Background] Hart B, Risley TR. Meaningful differences in the everyday experience of young American children. Baltimore, MD: Paul Brookes Publishing Company; 1995.
- [Background] Zuckerman B, Augustyn M. Books and reading: evidence-based standard of care whose time has come. Acad Pediatr. 2011 Jan-Feb;11(1):11-7. doi: 10.1016/j.acap.2010.09.007. PMID 21272819
- [Background] Payne AC, Whitehurst GJ, Angell aL. The role of home literacy environment in the development of language ability in preschool children from low-income families. Early Child Res Q. 1994:427-440.
- [Background] Weinberger J. A longitudinal study of children's early literacy experiences at home and later literacy development at home and school. J Res Reading. 1996;19:14-24.
- [Background] Senechal M, Lefevre J, Thomas EM, Daley KE. Differential effects of home literacy experiences on the development of oral and written language. Reading Res Q. 1998;33:96-116.
- [Background] Jimenez ME, Mendelsohn AL, Lin Y, Shelton P, Reichman N. Early Shared Reading Is Associated with Less Harsh Parenting. J Dev Behav Pediatr. 2019 Sep;40(7):530-537. doi: 10.1097/DBP.0000000000000687. PMID 31107765
- [Background] Jimenez ME, Hudson SV, Lima D, Mendelsohn AL, Pellerano M, Crabtree BF. Perspectives on shared reading among a sample of Latino parents. Child Care Health Dev. 2019 Mar;45(2):292-299. doi: 10.1111/cch.12634. Epub 2018 Dec 19. PMID 30471139
- [Background] Mendelsohn AL, Mogilner LN, Dreyer BP, Forman JA, Weinstein SC, Broderick M, Cheng KJ, Magloire T, Moore T, Napier C. The impact of a clinic-based literacy intervention on language development in inner-city preschool children. Pediatrics. 2001 Jan;107(1):130-4. doi: 10.1542/peds.107.1.130. PMID 11134446
- [Background] Asch DA, Muller RW, Volpp KG. Automated hovering in health care--watching over the 5000 hours. N Engl J Med. 2012 Jul 5;367(1):1-3. doi: 10.1056/NEJMp1203869. Epub 2012 Jun 20. No abstract available. PMID 22716935
- [Background] Whittaker R, McRobbie H, Bullen C, Rodgers A, Gu Y, Dobson R. Mobile phone text messaging and app-based interventions for smoking cessation. Cochrane Database Syst Rev. 2019 Oct 22;10(10):CD006611. doi: 10.1002/14651858.CD006611.pub5. PMID 31638271
- [Background] Jacobson Vann JC, Jacobson RM, Coyne-Beasley T, Asafu-Adjei JK, Szilagyi PG. Patient reminder and recall interventions to improve immunization rates. Cochrane Database Syst Rev. 2018 Jan 18;1(1):CD003941. doi: 10.1002/14651858.CD003941.pub3. PMID 29342498
- [Background] Taveras EM, Marshall R, Sharifi M, Avalon E, Fiechtner L, Horan C, Gerber MW, Orav EJ, Price SN, Sequist T, Slater D. Comparative Effectiveness of Clinical-Community Childhood Obesity Interventions: A Randomized Clinical Trial. JAMA Pediatr. 2017 Aug 7;171(8):e171325. doi: 10.1001/jamapediatrics.2017.1325. Epub 2017 Aug 7. PMID 28586856
- [Background] Ladley A, Hieger AW, Arthur J, Broom M. Educational Text Messages Decreased Emergency Department Utilization Among Infant Caregivers: A Randomized Trial. Acad Pediatr. 2018 Aug;18(6):636-641. doi: 10.1016/j.acap.2018.02.003. Epub 2018 Feb 9. PMID 29432907
- [Background] O'Leary ST, Lee M, Lockhart S, et al. Effectiveness and Cost of Bidirectional Text Messaging for Adolescent Vaccines and Well Care. Pediatrics. 2015;136(5):e20151089. Pediatrics. 2016 Sep;138(3):e20161768. doi: 10.1542/peds.2016-1768. No abstract available. PMID 27581853
- [Background] NICHD Strategic Plan 2020. NIH Pub Number 19-HD-8091. Bethesda, MD: Eunice Kennedy Shriver National Institute of Child Health and Human Development;2019.
- [Background] Dreyer BP, Mendelsohn AL, Tamis-LeMonda CS. Assessing the child's cognitive home environment through parental report: reliability and validity. Early Dev Parent. 1996;5:271-287.
- [Background] Reitman D, Currier RO, Stickle TR. A critical evaluation of the Parenting Stress Index-Short Form (PSI-SF) in a head start population. J Clin Child Adolesc Psychol. 2002 Sep;31(3):384-92. doi: 10.1207/S15374424JCCP3103_10. PMID 12149976
- [Background] Powell G, Mackrain M, LeBuffe P. Devereux Early Childhood Assessment for Infants and Toddlers- Technical Manual. Lewisville, NC: Kaplan Early Learning Corporation;2007.
- [Background] Feldman HM, Dollaghan CA, Campbell TF, Kurs-Lasky M, Janosky JE, Paradise JL. Measurement properties of the MacArthur communicative development inventories at ages one and two years. Child Dev. 2000 Mar-Apr;71(2):310-22. doi: 10.1111/1467-8624.00146. PMID 10834466

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants in phase 1were parents only and were enrolled between November 17, 2020-June 30,2022 at the two participating practices. Study participants in phase 2 were parent-child dyads and were enrolled from July 20, 2021-October 28, 2021 at the two participating practices.
Pre-assignment Details: 10 mothers of eligible children were enrolled in phase 1 and completed brief rapid cycle interviews. Demographic characteristics of these 10 participants were not collected.
Groups:
- Phase 1: consists of rapid cycle interviews
- Phase 2 Texting Arm: Text Messaging Only: Consist of daily text messages on shared reading
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
- Phase 2 Regret Arm: Text Messaging + Coaching: Will consist of Group 1 plus personalized coaching.
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
  Coaching: Personalized coaching content will be made available to participants through links in the text messages and will provide comparisons of their reading frequency with that of other participants.
- Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery: Will consist of Group 2 plus availability of a weekly lottery.
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
  Coaching: Personalized coaching content will be made available to participants through links in the text messages and will provide comparisons of their reading frequency with that of other participants.
  Lottery: Participants who reply to a text message that they read on a particular day will be entered into daily and weekly drawings to receive cash payments.
Period: Rapid Cycle Interviews (Phase 1)
Arm/Group | Phase 1 | Phase 2 Texting Arm: Text Messaging Only | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Started (Note: For phase 1, 10 mothers of eligible children were enrolled.) | 10 | 0 | 0 | 0
Completed (10 mothers completed Rapid Cycle Interviews) | 10 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0
Period: Randomized Controlled Trial (Phase 2)
Arm/Group | Phase 1 | Phase 2 Texting Arm: Text Messaging Only | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Started (For phase 2, dyads consisting of a single parent and eligible child were enrolled both virtually and in-person at 2 outpatient clinics.) | 0 | 15 | 15 | 15
Baseline Visit (45 Parent-child dyads completed baseline measures prior to randomization assignment) | 0 | 15 | 15 | 15
Completed (40 Parent-child dyads completed 2 month follow-up surveys) | 0 | 14 | 12 | 14
Not Completed | 0 | 1 | 3 | 1
Not completed — Lost to Follow-up | 0 | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: For phase 1, baseline characteristics of mothers participating in phase 1 rapid cycle interviews was not collected. In phase 2, a total of 43 Baseline measures were completed. Two participants did not complete the demographic survey measures (both in regret arm). A total of 3 participant did complete the StimQ-Read and PSI-SF at baseline (1 in control, 1 in regret and 1 in lottery arm).
Groups:
- Phase 2 Texting Arm: Text Messaging: Consist of daily text messages on shared reading
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
- Total: Total of all reporting groups
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery | Total
Number analyzed (Participants) | 15 | 15 | 15 | 45
Age, Continuous [Mean (Standard Deviation); unit: Months] — Demographic survey measure. Population: Age of child at enrollment (months), mean and SD provided.
  Months | 11.6 (4.7) | 11.9 (3.3) | 12.1 (4.2) | 11.8 (4.0)
Age, Continuous [Mean (Standard Deviation); unit: Years] — Demographic survey measure. Age of caregiver at enrollment (years), mean and SD provided.
  Years | 29.5 (6.7) | 24.8 (4.9) | 28.2 (3.9) | 27.6 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Demographic survey measure. Population: Sex of all participants enrolled in phase 2.
  Participants
    Sex of child enrolled: Female | 8 | 8 | 4 | 20
    Sex of child enrolled: Male | 7 | 7 | 11 | 25
    Sex of caregiver enrolled: Female | 14 | 13 | 15 | 42
    Sex of caregiver enrolled: Male | 1 | 2 | 0 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Demographic survey measure. Population: Characteristic of Ethnicity (n=43) for both child and caregiver enrolled in phase 2. A total of two participants did not complete measure.
  Participants
    Ethnicity of Children Enrolled: number analyzed (Participants) | 15 | 13 | 15 | 43
    Ethnicity of Children Enrolled: Hispanic or Latino | 1 | 0 | 1 | 2
    Ethnicity of Children Enrolled: Not Hispanic or Latino | 14 | 13 | 14 | 41
    Ethnicity of Children Enrolled: Unknown or Not Reported | 0 | 0 | 0 | 0
    Ethnicity of Caregiver Enrolled: number analyzed (Participants) | 15 | 13 | 15 | 43
    Ethnicity of Caregiver Enrolled: Hispanic or Latino | 1 | 0 | 1 | 2
    Ethnicity of Caregiver Enrolled: Not Hispanic or Latino | 14 | 13 | 14 | 41
    Ethnicity of Caregiver Enrolled: Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Demographic survey measure. Population: Race of child and caregiver enrolled in phase 2 of study. A total of two participants did not complete measure.
  Participants
    Child: number analyzed (Participants) | 15 | 13 | 15 | 43
    Child: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Child: Asian | 0 | 0 | 0 | 0
    Child: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Child: Black or African American | 14 | 8 | 13 | 35
    Child: White | 1 | 0 | 2 | 3
    Child: More than one race | 0 | 5 | 0 | 5
    Child: Unknown or Not Reported | 0 | 0 | 0 | 0
    Caregiver: number analyzed (Participants) | 15 | 13 | 15 | 43
    Caregiver: American Indian or Alaska Native | 0 | 0 | 0 | 0
    Caregiver: Asian | 0 | 0 | 0 | 0
    Caregiver: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Caregiver: Black or African American | 13 | 8 | 14 | 35
    Caregiver: White | 1 | 0 | 0 | 1
    Caregiver: More than one race | 1 | 5 | 1 | 7
    Caregiver: Unknown or Not Reported | 0 | 0 | 0 | 0
Recruitment Site [Count of Participants; unit: Participants] — Demographic survey measure.
  Participants
    Cobbs Creek | 3 | 2 | 1 | 6
    Karabots | 12 | 13 | 14 | 39
Children per caregiver [Mean (Standard Deviation); unit: avg. number children per caregiver] — Demographic survey measure. Number of children (mean) living at home with caregiver at time of enrollment. Population: A total of two participants did not complete measure.
  avg. number children per caregiver
    number analyzed (Participants) | 15 | 13 | 15 | 43
    (all) | 2.3 (1.8) | 1.8 (1.2) | 2.2 (1.1) | 2.1 (1.4)
Marital Status [Count of Participants; unit: Participants] — Demographic survey measure. Population: Marital status of caregivers enrolled in phase 2. A total of two participants (both in regret arm) did not complete measure.
  Participants
    number analyzed (Participants) | 15 | 13 | 15 | 43
    Married/Living together | 6 | 5 | 4 | 15
    Single, never married | 9 | 8 | 11 | 28
Education [Count of Participants; unit: Participants] — Demographic survey measure. Population: Education level of caregivers enrolled in phase 2. A total of two participant (both in regret arm) did not complete measure.
  Participants
    number analyzed (Participants) | 15 | 13 | 15 | 43
    Grades 9-11 | 0 | 2 | 1 | 3
    High School/GED | 6 | 5 | 10 | 21
    Some college/ college graduate | 9 | 5 | 3 | 17
    Post-college | 0 | 1 | 1 | 2
Income [Count of Participants; unit: Participants] — Demographic survey measure. Population: Income of caregivers enrolled in phase (n=37) 2. A total of 2 participants did not complete the measure and a total of 6 participants missing (chose not to answer).
  Participants
    number analyzed (Participants) | 13 | 12 | 12 | 37
    <$25,000 | 4 | 7 | 8 | 19
    $25,000 - $54,999 | 7 | 3 | 3 | 13
    >$55,000 | 2 | 2 | 1 | 5
Measure of Cognitive Stimulation Provided in the Home (Reading Subscale) [Mean (Standard Deviation); unit: units on a scale] — The Read subscale of the Measure of Cognitive Stimulation Provided in the Home (StimQ-read) is a validated 14-item parent self-report questionnaire designed to measure the home reading environment for children ages 5 to 72 months of age. The total score on the StimQ reading subscale will be used to assess changes in the child's reading environment from baseline to follow-up (2 months).
  Scores can range from a minimum score of 2 and a maximum score of 18 with a higher score indicating a better at home reading environment. Population: A total of 3 participants did not complete the StimQ-read measure at baseline.
  units on a scale
    number analyzed (Participants) | 14 | 14 | 14 | 42
    (all) | 12.9 (3.2) | 12.8 (4.5) | 15 (3.6) | 13.6 (3.8)
Parenting Stress Index-Short Form (PSI-SF) [Mean (Standard Deviation); unit: units on a scale] — The Parenting Stress Index-Short Form (PSI-SF) is a validated 36-item scale that measures parenting stress. Its been shown to have excellent internal consistency and to be positively associated with maternal psychological distress. Scores on the PSI-SF correlate well with the full PSI. It yields a Total Stress score from three scales: Parental Distress, Parent-Child Dysfunctional Interaction, and Difficult Child. The total score is used(range: 36-180), with higher scores indicating higher levels of stress. This measure will assess changes in PSI-SF from baseline to follow-up (2 months). Population: A total of 3 participants did not complete the PSI-SF measure at baseline.
  units on a scale
    number analyzed (Participants) | 14 | 14 | 14 | 42
    (all) | 56.3 (18.6) | 62.6 (22.5) | 53.6 (13.3) | 57.5 (18.5)

OUTCOME MEASURES:

1. Primary Outcome: Acceptability Survey
Description: To determine acceptability, participants will be assessed on their overall satisfaction (5-point Likert scale 1=strong disagree, 2=disagree, 3=not sure, 4=agree and 5= strongly agree) with the study delivery intervention and answered survey questions regarding likes and dislikes concerning the intervention group they received following the intervention period.
Time Frame: 2 months
Population: A total of 42 participant completed the measure. 3 participants were lost to follow-up
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 14 | 13 | 15
score on a scale | 4 (1.1) | 3.3 (1.3) | 3.8 (1.2)

2. Primary Outcome: Feasibility of Study
Description: Percentage of study participants who completed the 2-month follow-up
Time Frame: 2 months
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2 Texting Arm: Text Messaging Only | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery | Phase 1
Number analyzed (Participants) | 15 | 15 | 15 | 10
Participants | 14 | 13 | 15 | 10

3. Secondary Outcome: Change in Score of Cognitive Stimulation Provided in the Home Measure - (StimQ-Read)
Description: To determine change in home reading environment, Investigators will examine differences in the Read subscale of the measure of Cognitive Stimulation provided in the home (StimQ) from baseline to 2 months. The Read subscale of the StimQ is a validated 14-item parent self-report questionnaire designed to measure of the home reading environment for children ages 5 to 72 months of age with a maximum score of 18 and a minimum score of 0. The higher score indicates a better home reading environment. The change in score from baseline to follow-up (2-months) will be used.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 13 | 13 | 14
score on a scale | 1.8 (2.8) | 3.2 (4.0) | 1.3 (2.7)
Statistical Analysis 1: Comparison: Phase 2 Texting Arm: Text Messaging vs Phase 2 Regret Arm: Text Messaging + Coaching vs Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery; Analysis of Variance statistical testing; Test type: Superiority; p = 0.32, ANOVA; F-Statistic = 1.18

4. Secondary Outcome: Change in Score for The Parenting Stress Index - Short Form (PSI-SF)
Description: To determine change in parenting stress, Investigators will examine differences in the Parenting Stress Index- Short Form (PSI-SF) from baseline to follow-up (2 months). The PSI-SF is a validated 36-item scale that measures parenting stress, and it has been shown to have excellent internal consistency and to be positively associated with maternal psychological distress. The scores can range from 36 to 180 with an higher scores overall indicating higher levels of parenting stress. The change in score from baseline to follow-up (2-months) will be used.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 13 | 13 | 14
score on a scale | 2.2 (18.2) | 5.3 (16.4) | 9 (34.5)
Statistical Analysis 1: Comparison: Phase 2 Texting Arm: Text Messaging vs Phase 2 Regret Arm: Text Messaging + Coaching vs Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery; Test type: Superiority; p = 0.78, ANOVA; F-Statistic = 0.25

5. Secondary Outcome: Change in Weekly Parent-Child Shared Reading Frequency
Description: Investigators will measure reading frequency as the average number of days per week of reported parent-child shared reading.
  This is a measure of parent's self-reported reading frequency using question 2 from Cognitive Stimulation Provided in the Home Measure Reading Subscales, Parents are asked "How many days each week do you read children's books to your child?". Scores will be collected at baseline and at the 2-month follow-up. Change in reading frequency will be computed by subtracting the days reading at baseline from the days reading at follow-up.
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: days per week reading
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 14 | 13 | 15
days per week reading
  Days per week reading at baseline | 4.1 (1.8) | 4.0 (1.8) | 4.8 (1.5)
  Days per week reading at 2-month follow-up | 3.9 (2.0) | 4.2 (1.7) | 4.9 (1.5)
  Change in reading frequency (days per week | -0.3 (2.2) | 0.2 (2.6) | 0.1 (1.7)
Statistical Analysis 1: Comparison: Phase 2 Texting Arm: Text Messaging vs Phase 2 Regret Arm: Text Messaging + Coaching vs Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery; Test type: Superiority; p = 0.19, ANOVA

6. Secondary Outcome: Measure of Child Socio-Emotional Development Using Devereux Early Childhood Assessment (DECA)
Description: Investigators will measure child socio-emotional development at 2 months using the Devereax Early Childhood Assessment (DECA), a validated 33-item parent report of social emotional problems for children 9-36 months of age. All 33 items are used to calculate the raw total protective factor (TPF). 18/33 items are used to calculate raw Initiative sub scale (infant's ability to use independent thought and action to meet his/her needs). 15/33 items are used to calculate raw Attachment/Relationships sub scale (mutual, strong, long-lasting relationship between the infant and significant adults such as family members, and teachers). Higher scores indicate greater social emotional development.
  For all 33 items parents can report (Never 0, Rarely 1, Occasionally 2, Frequently 3, Very Frequently 4). Raw total scores can range from 0-132, with higher scores indicating a better outcome.
Time Frame: 2 months
Population: A total of 7 participants did not complete DECA. 3 participants were lost to follow-up and 4 participant scores were dropped (>18 mo at time of measure completion).
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Control: Text Messaging: Consist of daily text messages on shared reading
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
- Regret Arm: Text Messaging + Coaching: Will consist of Group 1 plus personalized coaching.
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
  Coaching: Personalized coaching content will be made available to participants through links in the text messages and will provide comparisons of their reading frequency with that of other participants.
- Lottery Arm: Text Messaging + Coaching + Lottery: Will consist of Group 2 plus availability of a weekly lottery.
  Text Messaging: Text Messages will be sent to participants using Penn's Way to Health Platform. Participants will be asked to reply to daily text messages on daily shared reading activities including the titles of books and time spent reading.
  Coaching: Personalized coaching content will be made available to participants through links in the text messages and will provide comparisons of their reading frequency with that of other participants.
  Lottery: Participants who reply to a text message that they read on a particular day will be entered into daily and weekly drawings to receive cash payments.
Arm/Group | Control: Text Messaging | Regret Arm: Text Messaging + Coaching | Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 13 | 12 | 13
score on a scale
  Initiative Score | 77.6 (18.7) | 64.3 (27.3) | 72.1 (28.6)
  Attachment/Relationship Score | 79.4 (19.4) | 66.6 (31.2) | 75.6 (27.8)
Statistical Analysis 1: Comparison: Control: Text Messaging vs Regret Arm: Text Messaging + Coaching vs Lottery Arm: Text Messaging + Coaching + Lottery; Test type: Superiority; p = 0.46, ANOVA

7. Secondary Outcome: Measure of Child Language Development Using MacArthur Communicative Development Inventory (CDI) - Percentiles
Description: Investigators measured child language development at 2 months using the MacArthur Communicative Development Inventory (CDI), a validated parent report scale of early child language development for children 8-30 months of age. Parents are asked to indicate the words their child understands but does not yet say in the first column (understands). For words that their child understands, Parents are asked to indicate which words their child says in the second column (understand and says).
  The raw total scores are inputted into a norming table for the CDI where a production (understand and says) and comprehension (understands) scores are generated based on the child's age and gender. Total scores can range from (0-178) with higher scores on the norming chart correlating to a higher percentile in comprehension or production. Total score is calculated by using summed scores where: blank = 0, understands = 1 and understands and speaks=2. Total scores were converted to percentile scores.
Time Frame: 2 months
Population: A total of 7 participants were unable to be used in CDI calculations. 3 participants were lost to follow-up and an additional 4 participant scores were dropped due to aging out of measure's age range (>18 mo at time survey was completed).
Measure: Mean (Standard Deviation); unit: Score Percentiles (%)
Arm/Group | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
Number analyzed (Participants) | 14 | 12 | 13
Score Percentiles (%) | 84.6 (29.7) | 78.5 (33.2) | 63.1 (42.6)
Statistical Analysis 1: Comparison: Phase 2 Texting Arm: Text Messaging vs Phase 2 Regret Arm: Text Messaging + Coaching vs Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery; Test type: Superiority; p = 0.30, ANOVA

ADVERSE EVENTS:
Time Frame: 1 year, 3 months
Groups:
- Phase 1: Rapid Cycle Interviews: Consists of a single instance of a rapid cycle interview
Arm/Group | Phase 1: Rapid Cycle Interviews | Phase 2 Texting Arm: Text Messaging | Phase 2 Regret Arm: Text Messaging + Coaching | Phase 2 Lottery Arm: Text Messaging + Coaching + Lottery
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/10 | 0/15 | 0/15 | 0/15

LIMITATIONS AND CAVEATS:
* Technical issues with W2H system: Group 2 texts that provided comparisons of participant reading frequency with that of other participant did not work properly for duration of study.
* Problem with Measurements leading to lost data:

  * CDI & DECA: data lost for participants >18 mo at follow-up visit
  * CDI: technical problems with RedCap data collection. Comprehension scores are uninterpretable. Only production scores were used in data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-04): https://cdn.clinicaltrials.gov/large-docs/81/NCT04576481/Prot_SAP_000.pdf